CLINICAL TRIAL: NCT03143790
Title: Ekstracorporal Shock Wave Therapy as a Treatment for Erectile Dysfunction in Men After Prostatectomy
Acronym: ESWT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Capacity problems
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martha Haahr M.D, M.D, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OUHL14.1
Record Dates: First submitted 2014-08-07; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Erectile Function
Keywords: Erectile Function; Prostatectomy; Extracorporeal Shock Wave Therapy; IIEF-5

STUDY DESIGN:
Intervention Model Description: Randomization to active or placebo treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient and therapist are blind. Primary investigator is not blind. Unblinding occurs 3 months after the end of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT (Active Comparator): 500 shockwave 3 different points on penis bilateral
  Interventions: Procedure: Extracorporeal Shockwave Terapy
- Placebo (Placebo Comparator): 500 shockwave 3 different points on penis bilateral
  Interventions: Procedure: Extracorporeal Shockwave Terapy

INTERVENTIONS:
Procedure: Extracorporeal Shockwave Terapy — Intervention is treatment with ESWT. Placebo treatment is using the same device as the active treatment, but the shock waves stopped in a non pressure-conductive filter
  Other Names: ESWT

SUMMARY:
Extra Corporal Shock wave Therapy Has proven effective as treatment with mild to moderate erectile dysfunction in men with erectile dysfunction. Investigator will examine whether the treatment also applies to men with moderate to severe erectile dysfunction after nerve injury associated with prostatectomy.

DETAILED DESCRIPTION:
All patients have undergone prostatectomy and are without recurrence. None of the men have sufficient effect of medical treatment for erectile dysfunction (tablets or injection therapy).

Each participant will fill out two validated sexual function questionnaires: IIEF-5 (International Index of Erectile Function), and EHS (Erection Hardness Score).

Our treatment protocol consists of one treatment sessions per week for 5 wk. The shockwaves are delivered to the distal, mid, and proximal penile shaft, and the left and right crura. The duration of each LI-ESWT session was about 20min, and each session comprised 500 shocks per treatment point (3000 per session) at an energy density of 0.15 mJ/mm2.

Patients are randomized to active treatment or placebo.By placebo added a blocking membrane in the machine, handling is carried out exactly the same way as the active treatment. None of the attending staff members will be familiar with who receive active and who receive placebo treatment.

For evaluation, the International index of erectile function (IIEF-5) will be used after 1, 3- and 6-mo follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Erectil dysfunction after radical prostatectomy less than two years ago
* IIEF - less than 20
* EHS - less than 4

Exclusion Criteria:

* drop out
* not sexual active
* penile prostesis

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only humans with a penis
Enrollment: 18 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 point | 1, 3 and 6 months
  Change in IIEF-5 point

CONTACTS AND LOCATIONS:
Locations (1):
- OUH, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
All results will be published